CLINICAL TRIAL: NCT00878332
Title: "Sandwich Osteotomy" Histologic Evaluation
Brief Title: Histologic Evaluation of Bone Formation After Alveolar Augmentation by "Sandwich Osteotomy" Procedure for Dental Implants Insertion
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Nardy Caspi, Hadassah medical center
Other Study IDs: sandwich osteotomy-HMO-CTIL
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2009-04-08 (Estimated); Status verified 2009-03

CONDITIONS: Dental Implants
Keywords: edentulous; fixed dental rehabilitation; insufficient bone height; Partially edentulous patients; Patients interested in fixed non removable dental rehabilitation by dental implants.; The recipient bone with insufficient bone height for dental implant insertion.; Adult patients
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Histologic slides
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- partially edentulous patients: Adult (post growth period) patients who are interested in fixed dental rehabilitation (non- removable denture) by dental implants.
  Partially edentulous patients with insufficient bone height for dental implant insertion.

SUMMARY:
The purpose of this study is to evaluate histologic bone remodeling after interpositional bone graft ("sandwich osteotomy" technique) using xenograft to fill the gap of the bone after moving and fixation it in the proper place.

DETAILED DESCRIPTION:
Dental implant use for partially edentolous jaw is a predictable procedure with high success rate. However, implantation procedure requires sufficient bone support both vertically and horizontally, and sometimes there is bone defect that requires bone augmentation prior to dental implant insertion.

There are some bone augmentation techniques known and used for this purposes, including: guided bone regeneration (GBR), distraction osteogenesis, split osteotomy, onlay bone graft, and interpositional bone graft.

One of the techniques is the interpositional bone graft using "sandwich osteotomy" technique, in which a cut is made in the bone (one horizontal and two vertical) separating a mobile bone portion which is fixed (using bone plate) in its new "ideal" position. The gap between the moved bone and the remaining bone is filled with xenograft ("bio-oss"). There is no documentation in the literature about histological evaluation of the bone after this well known clinical procedure. Four months after the bone augmentation procedure - the fixating plate is moved out and dental implants inserted. The first bur of the implantation (the smallest in the diameter) will be a trephine from which a histologic slide will be taken for check. The continuous dental implants insertion is the normal protocol for dental implantation (widening the recipient hole with bur, and insertion of the implant), followed by rehabilitation by prosthodontics.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* partially edentulous patients
* insufficient bone height (recipient site)
* interested in fixed dental rehabilitation using dental implants

Exclusion Criteria:

* smoking
* unbalanced diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients refered to the oral and maxillofacial clinic for bone augmentation (because of insufficient bone height) and fixed rehabilitation using dental implants
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Histologic slide evaluation of the bone on the dental implantation time | implantation day (four months post bone augmentation)

CONTACTS AND LOCATIONS:
Overall Officials: Nardy Caspi, MD / DMD, Principal Investigator — Senior Lecturer oral and maxillofacial surgery
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Jensen OT. Alveolar segmental "sandwich" osteotomies for posterior edentulous mandibular sites for dental implants. J Oral Maxillofac Surg. 2006 Mar;64(3):471-5. doi: 10.1016/j.joms.2005.11.030. PMID 16487811
- [Background] Jensen OT, Kuhlke L, Bedard JF, White D. Alveolar segmental sandwich osteotomy for anterior maxillary vertical augmentation prior to implant placement. J Oral Maxillofac Surg. 2006 Feb;64(2):290-6. doi: 10.1016/j.joms.2005.10.021. PMID 16413903
- [Background] Stellingsma C, Raghoebar GM, Meijer HJ, Batenburg RH. Reconstruction of the extremely resorbed mandible with interposed bone grafts and placement of endosseous implants. A preliminary report on outcome of treatment and patients' satisfaction. Br J Oral Maxillofac Surg. 1998 Aug;36(4):290-5. doi: 10.1016/s0266-4356(98)90713-6. PMID 9762457
- [Background] Marchetti C, Trasarti S, Corinaldesi G, Felice P. Interpositional bone grafts in the posterior mandibular region: a report on six patients. Int J Periodontics Restorative Dent. 2007 Dec;27(6):547-55. PMID 18092449
- [Background] Yeung R. Surgical management of the partially edentulous atrophic mandibular ridge using a modified sandwich osteotomy: a case report. Int J Oral Maxillofac Implants. 2005 Sep-Oct;20(5):799-803. PMID 16274157
- [Background] Robiony M, Costa F, Politi M. Alveolar sandwich osteotomy of the anterior maxilla. J Oral Maxillofac Surg. 2006 Sep;64(9):1453-4; author reply 1454-5. doi: 10.1016/j.joms.2006.02.006. No abstract available. PMID 16916686
- [Background] Politi M, Robiony M. Localized alveolar sandwich osteotomy for vertical augmentation of the anterior maxilla. J Oral Maxillofac Surg. 1999 Nov;57(11):1380-2. doi: 10.1016/s0278-2391(99)90883-2. No abstract available. PMID 10555808